CLINICAL TRIAL: NCT07058285
Title: Steps Against the Burden of Parkinson's Disease
Brief Title: Steps Against the Burden of Parkinson's Disease - RCT Kiel
Acronym: StepuP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Walter Maetzler, Prof. Dr., University of Kiel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6ef2e427b002
Record Dates: First submitted 2025-03-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Fall
Keywords: EEG; EMG; perturbation; daily-life gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiel (Experimental): In Kiel, the experimental group will engage in 12-sessions of SDTT with additional anteroposterior perturbations, contrasting with the control group undergoing regular SDTT.
  Interventions: Other: SDTT+ anteroposterior perturbations
- Control (Active Comparator)
  Interventions: Other: Speed-dependent treadmill training (SDTT)

INTERVENTIONS:
Other: Speed-dependent treadmill training (SDTT) — This training methodology focuses on adjusting the treadmill's speed according to the individual's walking pace, creating a more dynamic and adaptive exercise environment. SDTT is designed to mimic real-world walking conditions and challenges, promoting neuromuscular coordination, balance, and overall mobility. By tailoring the treadmill speed to match the user's gait, SDTT encourages the development of natural and efficient walking patterns. This training technique has shown promise in various clinical settings, aiding individuals with gait impairments caused by neurological conditions, musculoskeletal disorders, or post-injury rehabilitation. Its adaptability allows for progressive adjustments as a person's walking abilities improve, making it a versatile tool for optimizing gait mechanics and functional mobility. o ensure continued progress and integration into daily life, home-based walking training, supported by a phone application, will be included between T1 and T2.
  Arms: Control
Other: SDTT+ anteroposterior perturbations — The SDTT+ anteroposterior perturbations program will trigger reactive gait adaptations by accelerations and decelerations of one of the belts of a split-belt treadmill.
  Arms: Kiel

SUMMARY:
Parkinson's disease (PD) affects over 10 million worldwide, causing unstable gait and falls in 70% of patients despite medication. This leads to confidence loss, isolation, fractures, and hospitalizations. Treadmill training, augmented by mechanical/virtual-reality triggers, has proven effective in enhancing gait and reducing falls. However, underlying treadmill training mechanisms are unclear. To personalize training, we'll explore how PD patients benefit and transfer effects to daily life.

This trial is part of three parallel randomized controlled trials within the Steps Against the Burden of Parkinson's Disease (CT-IDs: 6ef2e427b002, 6ef2e427b003, 6ef2e427b004) project, which will perform a pooled analysis across all sites in addition to individual RCT analyses. Each trial adheres to a shared core protocol while allowing for adaptations in the perturbation protocol, ensuring that data can be combined. Importantly, mechanistic findings and outcomes from this specific RCT will be reported independently, but also as part of a pooled analysis.

In this trials, PD patients will undergo treadmill training with and without adaptations (perturbations). 12 sessions of treadmill training will be provided, with pre/post assessments and a Follow-up 12±2 weeks following T1 with pre/post assessments and a Follow-up 12±2 weeks following T1 at 8 to 12 weeks after the post assessment. For post treadmill training a phone app will be offered as a home-based speed dependent walk training intervention. This intervention is an App based training for gait adaptability and allows users to set their own training time and pace. It delivers a rhythmic metronomic beat for three different walking speeds, designed to trigger movement and encourage better walking patterns. Gait improvements are expected, driven by sensorimotor integration improving balance control. Biomechanical data analysis will reveal enhanced foot placement control. Neurophysiological changes will be studied through EEG and EMG, aiming to find improved gait stability with reduced EEG beta power and increased EEG-EMG coherence.

Gait improvement in the lab might not correlate with daily-life results. Gait self-efficacy could influence transfer, prompting investigation into mechanistic associations with mobility outcomes. Remote digital tools will assess week-long mobility outcomes, employing machine learning to comprehend why some improve both in lab and life, while others don't. This will uncover mechanisms translating treatment effects into real-world outcomes, aiding personalized intervention development.

DETAILED DESCRIPTION:
i. Rationale The rationale of this trial is that speed dependent treadmill training (SDTT) improves gait through improved sensorimotor integration, with changes in cortical activity as neural correlates. Additional benefits of treadmill training can be seen if perturbation or adaptations are added. This is based on the idea, that in addition to the sensorimotor integration the reactive balance in trained as well18. Furthermore, it hypothesizes that treadmill training and its effects on gait quality will improve gait self-efficacy, which mediates and/or modifies transfer of training effects to improved daily-life gait.

ii. Objectives

Thus, the objectives of our StepuP project are:

1. To understand the kinematic and neural mechanisms that underlie improvements in gait due to treadmill training with and without mechanically and VR-triggered gait adaptations in people with PD;
2. To assess to what extent improvements in gait due to treadmill training, as measured in the lab, transfer to improvements in daily life mobility;
3. To understand the mechanisms that underpin transfer from improvements in gait to improvements of mobility in daily life in people with PD;
4. To understand for whom treadmill training improves lab-based gait characteristics and for whom it does not, and understand for whom treadmill training improves mobility in daily life and for whom it does not.

Attaining these objectives will provide a better understanding of the successes and failures of treadmill training to improve gait stability and prevent falls in people with PD at an individual level, which in the medium term will allow targeted delivery of such interventions and in the long term will allow personalization of such interventions to improve outcomes for all.

iii. Endpoints Concerning the endpoints, this trial examines the effect of treadmill training with and without perturbations on gait performance, and neural correlates in people with PD. The primary endpoint is (change in) gait speed, secondary endpoints are divided into three groups (clinical, kinematic and neurophysiological). Clinical measures are used to assess the effect of training on disease symptoms. Kinematic measures are changes from baseline to Follow-up 12±2 weeks following T1, all under controlled conditions (treadmill), and provide insight into gait performance and quality. Neurophysiological measures aim to understand the neural control mechanisms underlying the training effects. On an exploratory level, the study aims to assess the training effects on daily-life gait by using wearable devices and assess gait self-efficacy using previously validated questionnaires.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of PD according to the MDS Criteria
2. Hoehn and Yahr stages I to III;
3. Movement Disorder Society-sponsored version of the Unified Parkinson Disease Rating Scale (MDS-UPDRS) gait sub-score of 1 or more
4. Signed informed consent to participation

Exclusion criteria

* Any known general health condition likely to interfere with or to pose a contraindication to non-medically supervised physical exercise.
* Moderate or severe depression (BDI-II ≥18)
* Cognitive impairment which may preclude the possibility to provide a fully informed consent to enrolment.
* Linguistic comprehension capacity less than 75% in ordinary conversation
* Severe psychiatric comorbidity which may interfere with compliance to the study protocol
* History of or current status of substance dependency
* Unable to walk less than 1 floor
* Thoracic pain in the last 4 weeks
* Currently enrolled in other interventional studies
* Implanted Deep Brain Stimulation device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Gait speed - T0 | Baseline
  Comfortable walking speed overground
Gait speed - T1 | After Intervention (2-12 weeks)
  Comfortable walking speed overground
Gait speed - T2 | After Follow-up 12±2 weeks following T1 (20-32 weeks)
  Comfortable walking speed overground

SECONDARY OUTCOMES:
Fall events (occurrence and frequency) and fall related injuries - T0 | Baseline (T0)
  The number of falls and whether the falls were injurious will be recorded. Twelve-month retrospective.
Fracture history - T0 | Baseline (T0)
  Number and type of fracture sustained will be recorded. Twelve-month retrospective.
Medication - T0 | Baseline (T0)
  Current medication will be recorded at each visit.
Medication - T1 | After Intervention (2-12 weeks)
  Current medication will be recorded at each visit.
Medication - T2 | Follow-up 12±2 weeks following T1
  Current medication will be recorded at each visit.
Euro-Quality of life (EQ-5D) - T0 | Baseline (T0)
  The first part is a descriptive system, assessing health in five dimensions.The second part of the questionnaire consists of a visual analog scale (VAS) on which patients mark their perceived level of health on a scale ranging from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
Euro-Quality of life (EQ-5D) - T1 | After Intervention (2-12 weeks)
  The first part is a descriptive system, assessing health in five dimensions.The second part of the questionnaire consists of a visual analog scale (VAS) on which patients mark their perceived level of health on a scale ranging from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
Euro-Quality of life (EQ-5D) - T2 | Follow-up 12±2 weeks following T1
  The first part is a descriptive system, assessing health in five dimensions.The second part of the questionnaire consists of a visual analog scale (VAS) on which patients mark their perceived level of health on a scale ranging from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
Frailty Index (FI) - T0 | Baseline (T0)
  Measures frailty based on five criteria: shrinking, low physical endurance/energy, low physical activity, weakness, and slow walking speed.
Frailty Index (FI) - T1 | After Intervention (2-12 weeks)
  Measures frailty based on five criteria: shrinking, low physical endurance/energy, low physical activity, weakness, and slow walking speed. For the Frailty Index, higher scores mean a worse outcome (increased frailty).
Frailty Index (FI) - T2 | Follow-up 12±2 weeks following T1
  Measures frailty based on five criteria: shrinking, low physical endurance/energy, low physical activity, weakness, and slow walking speed. For the Frailty Index, higher scores mean a worse outcome (increased frailty).
Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue scale - T0 | Baseline (T0)
  Measures fatigue during usual daily activities over the past week. The FACIT-F scale consists of 13 items, each scored from 0 (Not at all) to 4 (Very much). Some items are reverse-scored. The total score ranges from 0 to 52. For the FACIT-F scale, higher scores indicate less fatigue (a better outcome).
Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue scale - T1 | After Intervention (2-12 weeks)
  Measures fatigue during usual daily activities over the past week. The FACIT-F scale consists of 13 items, each scored from 0 (Not at all) to 4 (Very much). Some items are reverse-scored. The total score ranges from 0 to 52. For the FACIT-F scale, higher scores indicate less fatigue (a better outcome).
Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue scale - T2 | Follow-up 12±2 weeks following T1
  Measures fatigue during usual daily activities over the past week. The FACIT-F scale consists of 13 items, each scored from 0 (Not at all) to 4 (Very much). Some items are reverse-scored. The total score ranges from 0 to 52. For the FACIT-F scale, higher scores indicate less fatigue (a better outcome).
Kinematics: 3D motion capture data - T0 | Baseline
  3D motion capture data.
Kinematics: 3D motion capture data - T1 | After Intervention (2-12 weeks)
  3D motion capture data.
Kinematics: 3D motion capture data - T2 | Follow-up 12±2 weeks following T1
  3D motion capture data.
Electroencephalography (EEG) - T0 | Baseline
  EEG measures brain activity to assess cortical involvement and sensorimotor integration for foot placement control. We'll specifically analyze beta power and beta band corticomuscular coherence with the rectus femoris muscle. Before analysis, EEG data will be cleaned using filtering and ICA to remove artifacts like muscle and eye movements. Coherence will be computed across the gait cycle using time-normalized EEG and EMG cross-spectra, and beamforming will localize sources.
Electroencephalography (EEG) - T1 | After Intervention (2-12 weeks)
  EEG measures brain activity to assess cortical involvement and sensorimotor integration for foot placement control. We'll specifically analyze beta power and beta band corticomuscular coherence with the rectus femoris muscle. Before analysis, EEG data will be cleaned using filtering and ICA to remove artifacts like muscle and eye movements. Coherence will be computed across the gait cycle using time-normalized EEG and EMG cross-spectra, and beamforming will localize sources.
Electroencephalography (EEG) - T2 | Follow-up 12±2 weeks following T1
  EEG measures brain activity to assess cortical involvement and sensorimotor integration for foot placement control. We'll specifically analyze beta power and beta band corticomuscular coherence with the rectus femoris muscle. Before analysis, EEG data will be cleaned using filtering and ICA to remove artifacts like muscle and eye movements. Coherence will be computed across the gait cycle using time-normalized EEG and EMG cross-spectra, and beamforming will localize sources.
Electromyography (EMG) - T0 | Baseline
  Surface EMG records electrical activity of superficial muscles to assess muscle function, fatigue, and activation patterns.
Electromyography (EMG) - T1 | After Intervention (2-12 weeks)
  Surface EMG records electrical activity of superficial muscles to assess muscle function, fatigue, and activation patterns.
Electromyography (EMG) - T2 | Follow-up 12±2 weeks following T1
  Surface EMG records electrical activity of superficial muscles to assess muscle function, fatigue, and activation patterns.
Gait speed (Preferred and maximal) - T0 | Baseline
  Preferred gait speed and maximal gait speed using a 20-m walk test will be derived.
Gait speed (Preferred and maximal) - T1 | After Intervention (2-12 weeks)
  Preferred gait speed and maximal gait speed using a 20-m walk test will be derived.
Gait speed (Preferred and maximal) - T2 | Follow-up 12±2 weeks following T1
  Preferred gait speed and maximal gait speed using a 20-m walk test will be derived.
Use of mobility aids - T0 | Baseline
  The use of commonly used walking aids (indoor and outdoor) will be recorded.
Use of mobility aids - T2 | Follow-up 12±2 weeks following T1
  The use of commonly used walking aids (indoor and outdoor) will be recorded.
Timed Up and Go (TUG) - T0 | Baseline
  A common clinical measure to assess mobility, balance, and walking ability in older adults.
Timed Up and Go (TUG) - T1 | After Intervention (2-12 weeks)
  A common clinical measure to assess mobility, balance, and walking ability in older adults.
Timed Up and Go (TUG) - T2 | Follow-up 12±2 weeks following T1
  A common clinical measure to assess mobility, balance, and walking ability in older adults.
Two-minute walking test (2MWT) - T0 | Baseline
  Measures functional exercise capacity. Distance in meters covered in 6 minutes is recorded.
Two-minute walking test (2MWT) - T1 | After Intervention (2-12 weeks)
  Measures functional exercise capacity. Distance in meters covered in 6 minutes is recorded.
Two-minute walking test (2MWT) - T2 | Follow-up 12±2 weeks following T1
  Measures functional exercise capacity. Distance in meters covered in 6 minutes is recorded.
Mini-BESTest - T0 | Baseline
  The Mini-BESTest (Mini-Balance Evaluation Systems Test) is a clinical balance assessment tool designed to evaluate various balance control systems. It assesses an individual's balance and stability on a series of functional tasks. The unabbreviated scale title is Mini-Balance Evaluation Systems Test (Mini-BESTest). It has a minimum value of 0 and a maximum value of 28. The Mini-BESTest is comprised of 14 items, each scored on a 3-point ordinal scale (0 = severe impairment, 1 = moderate impairment, 2 = no impairment). The scores from all items are summed to provide a total score. Higher scores on the Mini-BESTest indicate better balance and stability, representing a better outcome.
Mini-BESTest - T1 | After Intervention (2-12 weeks)
  The Mini-BESTest (Mini-Balance Evaluation Systems Test) is a clinical balance assessment tool designed to evaluate various balance control systems. It assesses an individual's balance and stability on a series of functional tasks. The unabbreviated scale title is Mini-Balance Evaluation Systems Test (Mini-BESTest). It has a minimum value of 0 and a maximum value of 28. The Mini-BESTest is comprised of 14 items, each scored on a 3-point ordinal scale (0 = severe impairment, 1 = moderate impairment, 2 = no impairment). The scores from all items are summed to provide a total score. Higher scores on the Mini-BESTest indicate better balance and stability, representing a better outcome.
Mini-BESTest - T2 | Follow-up 12±2 weeks following T1
  The Mini-BESTest (Mini-Balance Evaluation Systems Test) is a clinical balance assessment tool designed to evaluate various balance control systems. It assesses an individual's balance and stability on a series of functional tasks. The unabbreviated scale title is Mini-Balance Evaluation Systems Test (Mini-BESTest). It has a minimum value of 0 and a maximum value of 28. The Mini-BESTest is comprised of 14 items, each scored on a 3-point ordinal scale (0 = severe impairment, 1 = moderate impairment, 2 = no impairment). The scores from all items are summed to provide a total score. Higher scores on the Mini-BESTest indicate better balance and stability, representing a better outcome.
Modified Gait Efficacy Scale (mGES) - T0 | Baseline
  The Modified Gait Efficacy Scale (mGES) assesses an individual's confidence in their walking ability across various challenging everyday circumstances. It is a self-report measure. The unabbreviated scale title is Modified Gait Efficacy Scale (mGES). It has a minimum value of 0 and a maximum value of 100. The mGES typically consists of several items where individuals rate their confidence on a scale (e.g., 0-10 or 0-100) for various walking situations. The total score is often calculated as an average or sum and then converted to a percentage. Higher scores on the Modified Gait Efficacy Scale indicate greater walking confidence, representing a better outcome.
Modified Gait Efficacy Scale (mGES) - T1 | After Intervention (2-12 weeks)
  The Modified Gait Efficacy Scale (mGES) assesses an individual's confidence in their walking ability across various challenging everyday circumstances. It is a self-report measure. The unabbreviated scale title is Modified Gait Efficacy Scale (mGES). It has a minimum value of 0 and a maximum value of 100. The mGES typically consists of several items where individuals rate their confidence on a scale (e.g., 0-10 or 0-100) for various walking situations. The total score is often calculated as an average or sum and then converted to a percentage. Higher scores on the Modified Gait Efficacy Scale indicate greater walking confidence, representing a better outcome.
Modified Gait Efficacy Scale (mGES) - T2 | Follow-up 12±2 weeks following T1
  The Modified Gait Efficacy Scale (mGES) assesses an individual's confidence in their walking ability across various challenging everyday circumstances. It is a self-report measure. The unabbreviated scale title is Modified Gait Efficacy Scale (mGES). It has a minimum value of 0 and a maximum value of 100. The mGES typically consists of several items where individuals rate their confidence on a scale (e.g., 0-10 or 0-100) for various walking situations. The total score is often calculated as an average or sum and then converted to a percentage. Higher scores on the Modified Gait Efficacy Scale indicate greater walking confidence, representing a better outcome.
Hand grip strength - T0 | Baseline
  Hand grip strength.
Short Falls Efficacy Scale International (Short FES-i) - T0 | Baseline
  The Short Falls Efficacy Scale International (Short FES-I) measures the level of concern about falling during social and physical activities, both inside and outside the home. It is a widely used self-report questionnaire. It has a minimum value of 7 and a maximum value of 28. The Short FES-I consists of 7 items. Each item is rated on a 4-point scale, from 1 (not concerned at all) to 4 (completely concerned). The scores for all 7 items are summed. Higher scores on the Short FES-I indicate a greater concern about falling, representing a worse outcome.
Short Falls Efficacy Scale International (Short FES-i) - T1 | After Intervention (2-12 weeks)
  The Short Falls Efficacy Scale International (Short FES-I) measures the level of concern about falling during social and physical activities, both inside and outside the home. It is a widely used self-report questionnaire. It has a minimum value of 7 and a maximum value of 28. The Short FES-I consists of 7 items. Each item is rated on a 4-point scale, from 1 (not concerned at all) to 4 (completely concerned). The scores for all 7 items are summed. Higher scores on the Short FES-I indicate a greater concern about falling, representing a worse outcome.
Short Falls Efficacy Scale International (Short FES-i) - T2 | Follow-up 12±2 weeks following T1
  The Short Falls Efficacy Scale International (Short FES-I) measures the level of concern about falling during social and physical activities, both inside and outside the home. It is a widely used self-report questionnaire. It has a minimum value of 7 and a maximum value of 28. The Short FES-I consists of 7 items. Each item is rated on a 4-point scale, from 1 (not concerned at all) to 4 (completely concerned). The scores for all 7 items are summed. Higher scores on the Short FES-I indicate a greater concern about falling, representing a worse outcome.
Montreal Cognitive Assessment (MoCA) - T0 | Baseline
  The Montreal Cognitive Assessment (MoCA) is a quick screening tool designed to detect mild cognitive impairment, assessing a broad range of cognitive domains. It has a minimum value of 0 and a maximum value of 30. The MoCA assesses attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. Each correct response contributes to the total score. A score of 26 or above is generally considered normal. Higher scores on the MoCA indicate better cognitive function, representing a better outcome.
Montreal Cognitive Assessment (MoCA) - T2 | Follow-up 12±2 weeks following T1
  The Montreal Cognitive Assessment (MoCA) is a quick screening tool designed to detect mild cognitive impairment, assessing a broad range of cognitive domains. It has a minimum value of 0 and a maximum value of 30. The MoCA assesses attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. Each correct response contributes to the total score. A score of 26 or above is generally considered normal. Higher scores on the MoCA indicate better cognitive function, representing a better outcome.
Color Trail Test (CTT) - T0 | Baseline
  The Color Trail Test (CTT) is a neuropsychological assessment with two parts (CTT-1, CTT-2) that evaluates cognitive flexibility, visual scanning, and executive function. Participants connect numbered circles, then alternate between numbers and letters.
  Key measures are completion time (min 0s, max typically 120-240s) and errors. Lower times and fewer errors indicate better attention, mental flexibility, and processing speed, signifying a better outcome.
Color Trail Test (CTT) - T2 | Follow-up 12±2 weeks following T1
  The Color Trail Test (CTT) is a neuropsychological assessment with two parts (CTT-1, CTT-2) that evaluates cognitive flexibility, visual scanning, and executive function. Participants connect numbered circles, then alternate between numbers and letters.
  Key measures are completion time (min 0s, max typically 120-240s) and errors. Lower times and fewer errors indicate better attention, mental flexibility, and processing speed, signifying a better outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - T0 | Baseline
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive, clinician-rated scale used to assess the severity and progression of Parkinson's Disease. Part III specifically focuses on the Motor Examination. It has a minimum value of 0 and a maximum value of 132 (sum of all 33 items in Part III, each scored 0-4). Part III consists of 33 items (e.g., speech, facial expression, rigidity, tremor, bradykinesia, gait, postural stability), each scored from 0 (normal) to 4 (severe impairment). The scores for all items are summed. Higher scores on the MDS-UPDRS Part III indicate greater motor impairment and more severe Parkinson's disease symptoms, representing a worse outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - T1 | After Intervention (2-12 weeks)
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive, clinician-rated scale used to assess the severity and progression of Parkinson's Disease. Part III specifically focuses on the Motor Examination. It has a minimum value of 0 and a maximum value of 132 (sum of all 33 items in Part III, each scored 0-4). Part III consists of 33 items (e.g., speech, facial expression, rigidity, tremor, bradykinesia, gait, postural stability), each scored from 0 (normal) to 4 (severe impairment). The scores for all items are summed. Higher scores on the MDS-UPDRS Part III indicate greater motor impairment and more severe Parkinson's disease symptoms, representing a worse outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - T2 | Follow-up 12±2 weeks following T1
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive, clinician-rated scale used to assess the severity and progression of Parkinson's Disease. Part III specifically focuses on the Motor Examination. It has a minimum value of 0 and a maximum value of 132 (sum of all 33 items in Part III, each scored 0-4). Part III consists of 33 items (e.g., speech, facial expression, rigidity, tremor, bradykinesia, gait, postural stability), each scored from 0 (normal) to 4 (severe impairment). The scores for all items are summed. Higher scores on the MDS-UPDRS Part III indicate greater motor impairment and more severe Parkinson's disease symptoms, representing a worse outcome.
New Freezing of Gait Questionnaire (NFOGQ) - T0 | Baseline
  The New Freezing of Gait Questionnaire (NFOGQ) is a patient-reported outcome measure specifically designed to detect and evaluate the impact and severity of freezing of gait (FOG) in individuals with Parkinson's disease or other neurological conditions. It has a minimum value of 0 and a maximum value of 45. The NFOGQ consists of 9 items, with a total score calculated by summing the scores for all items. Each item is typically scored on a 5-point Likert scale. Higher scores on the NFOGQ indicate a greater severity, frequency, and impact of freezing of gait, representing a worse outcome.
New Freezing of Gait Questionnaire (NFOGQ) - T1 | After Intervention (2-12 weeks)
  The New Freezing of Gait Questionnaire (NFOGQ) is a patient-reported outcome measure specifically designed to detect and evaluate the impact and severity of freezing of gait (FOG) in individuals with Parkinson's disease or other neurological conditions. It has a minimum value of 0 and a maximum value of 45. The NFOGQ consists of 9 items, with a total score calculated by summing the scores for all items. Each item is typically scored on a 5-point Likert scale. Higher scores on the NFOGQ indicate a greater severity, frequency, and impact of freezing of gait, representing a worse outcome.
New Freezing of Gait Questionnaire (NFOGQ) - T2 | Follow-up 12±2 weeks following T1
  The New Freezing of Gait Questionnaire (NFOGQ) is a patient-reported outcome measure specifically designed to detect and evaluate the impact and severity of freezing of gait (FOG) in individuals with Parkinson's disease or other neurological conditions. It has a minimum value of 0 and a maximum value of 45. The NFOGQ consists of 9 items, with a total score calculated by summing the scores for all items. Each item is typically scored on a 5-point Likert scale. Higher scores on the NFOGQ indicate a greater severity, frequency, and impact of freezing of gait, representing a worse outcome.
Home assessment: Steps per day - T0 | Baseline (T0)
  The steps per day will be recorded.
Home assessment: Steps per day - T1 | After Intervention (2-12 weeks)
  The steps per day will be recorded.
Home assessment: Steps per day - T2 | Follow-up 12±2 weeks following T1
  The steps per day will be recorded.
Home assessment: Amount and length of uninterrupted walk durations - T0 | Baseline (T0)
  The amount and length of uninterrupted walk durations will be determined.
Home assessment: Amount and length of uninterrupted walk durations - T1 | After Intervention (2-12 weeks)
  The amount and length of uninterrupted walk durations will be determined.
Home assessment: Amount and length of uninterrupted walk durations - T2 | Follow-up 12±2 weeks following T1
  The amount and length of uninterrupted walk durations will be determined.
Home assessment: Stride time variability - T0 | Baseline (T0)
  The stride time variability will be derived.
Home assessment: Stride time variability - T1 | After Intervention (2-12 weeks)
  The stride time variability will be derived.
Home assessment: Stride time variability - T2 | Follow-up 12±2 weeks following T1
  The stride time variability will be derived.
Home assessment: Symmetry of gait - T0 | Baseline (T0)
  Symmetry of gait will be determined.
Home assessment: Symmetry of gait - T1 | After Intervention (2-12 weeks)
  Symmetry of gait will be determined.
Home assessment: Symmetry of gait - T2 | Follow-up 12±2 weeks following T1
  Symmetry of gait will be determined.
Home assessment: FOG episodes, Medication, and Physical activity (self-reports) - T0 | Baseline (T0)
  FOG episodes, Medication and Physical activity will be recorded by self-reports.
Home assessment: FOG episodes, Medication, and Physical activity (self-reports) - T1 | After Intervention (2-12 weeks)
  FOG episodes, Medication and Physical activity will be recorded by self-reports.
Home assessment: Weekly Calendars for Physical activity, Falls and Injurious Falls - T0 | Baseline (T0)
  Weekly Calendars will be used to assess Physical activity, Falls and Injurious Falls.
Home assessment: Weekly Calendars for Physical activity, Falls and Injurious Falls - T1 | After Intervention (2-12 weeks)
  Weekly Calendars will be used to assess Physical activity, Falls and Injurious Falls.
Home assessment: Weekly Calendars for Physical activity, Falls and Injurious Falls - T2 | Follow-up 12±2 weeks following T1
  Weekly Calendars will be used to assess Physical activity, Falls and Injurious Falls.
Acceptability and satisfaction with the intervention (System Usability Scale and PACES) - T1 | After Intervention (2-12 weeks)
  The Physical Activity Enjoyment Scale (PACES) is a self-report questionnaire designed to measure an individual's enjoyment of physical activity. It typically consists of 18 items where participants rate their feelings about physical activity on a 7-point bipolar scale. It has a minimum possible score of 18 (if each item is rated '1') and a maximum possible score of 126 (if each item is rated '7'). Scores from all 18 items are summed to create a total score. Higher scores on the PACES indicate greater enjoyment of physical activity, representing a better outcome. Additionally it includes questions developed specifically for the components of this study.
Acceptability and satisfaction with the intervention (System Usability Scale and PACES) - T2 | Follow-up 12±2 weeks following T1
  The Physical Activity Enjoyment Scale (PACES) is a self-report questionnaire designed to measure an individual's enjoyment of physical activity. It typically consists of 18 items where participants rate their feelings about physical activity on a 7-point bipolar scale. It has a minimum possible score of 18 (if each item is rated '1') and a maximum possible score of 126 (if each item is rated '7'). Scores from all 18 items are summed to create a total score. Higher scores on the PACES indicate greater enjoyment of physical activity, representing a better outcome. Additionally it includes questions developed specifically for the components of this study.
Changes in attitudes towards physical activity (Exercise Self-Efficacy Scale) - T1 | After Intervention (2-12 weeks)
  The Exercise Self-Efficacy Scale (ESES) is designed to assess an individual's confidence in their ability to engage in regular exercise, particularly in challenging situations. There are various versions of self-efficacy scales, but they generally follow a similar structure. It has a minimum possible score of 0 (or the lowest point on the chosen confidence scale) and a maximum possible score of 100 (or the highest point on the chosen confidence scale). Participants typically rate their confidence for various exercise-related scenarios on a percentage scale, for instance, 0% = not at all confident to 100% = completely confident. The scores are then averaged or summed. Higher scores on the Exercise Self-Efficacy Scale indicate greater confidence in one's ability to exercise, representing a better outcome.
Changes in attitudes towards physical activity (Exercise Self-Efficacy Scale) - T2 | Follow-up 12±2 weeks following T1
  The Exercise Self-Efficacy Scale (ESES) is designed to assess an individual's confidence in their ability to engage in regular exercise, particularly in challenging situations. There are various versions of self-efficacy scales, but they generally follow a similar structure. It has a minimum possible score of 0 (or the lowest point on the chosen confidence scale) and a maximum possible score of 100 (or the highest point on the chosen confidence scale). Participants typically rate their confidence for various exercise-related scenarios on a percentage scale, for instance, 0% = not at all confident to 100% = completely confident. The scores are then averaged or summed. Higher scores on the Exercise Self-Efficacy Scale indicate greater confidence in one's ability to exercise, representing a better outcome.
Exit interviews (Barriers and enablers to long-term use) - T1 | After Intervention (2-12 weeks)
  Exit interviews will be conducted to explore the barriers and enablers to long-term use and reasons for ceased involvement (if applicable) using pre-prepared, open-ended questions according to qualitative interview methods.
Exit interviews (Barriers and enablers to long-term use) - T2 | Follow-up 12±2 weeks following T1
  Exit interviews will be conducted to explore the barriers and enablers to long-term use and reasons for ceased involvement (if applicable) using pre-prepared, open-ended questions according to qualitative interview methods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
To ensure high standards of data curation, the widely accepted Brain Imaging Data Structure (BIDS) standard to store the motion, EMG and EEG data will be followed and data will be made public in a coded, de-identified manner.
Supporting Information: Study Protocol, Analytic Code